CLINICAL TRIAL: NCT05435196
Title: Efficacy of High-intensity Exercise in Women With Prediabetes: Randomized, Controlled Trial, With Six Months Followed
Brief Title: Efficacy of High-intensity Exercise in Women With Prediabetes
Acronym: Prediabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Popular Autónoma del Estado de Puebla (Other)
Collaborators: Hospital de Especialidades 5 de mayo, ISSSTEP. Puebla, México (Unknown); University of Alcala (Other)
Responsible Party: Principal Investigator, Clara Luz Pérez Quiroga, Clinical professor, Universidad Popular Autónoma del Estado de Puebla
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CLPQ
Record Dates: First submitted 2022-05-26; First posted 2022-06-28 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Prediabetic State
Keywords: prediabetic state; exercise therapy; women
MeSH Terms: conditions — Prediabetic State | interventions — Exercise Therapy; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: An initial evaluation, a final one, will be carried out 3 months and 6 months after the end of the study.
Who Masked: Investigator
Masking Description: Masking of the outcome variables
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Get the training in with high-intensity interval exercise. Will be applied through 10 sets of 60 seconds. The first 30 seconds will consist of going up and down a step 15 cm high, immediately 30 seconds of squats as fast as possible with 90° knee flexion. The recovery period between each set will be 60 seconds, with a low-intensity activity (light walking). Based on high-intensity exercise, we must achieve an effort greater than 85% of the maximum frequency, using the heart rate meter and its equivalences with the Perceived Effort Scale (RPE).
  Receive a multimodal training that will consist of: resistance exercises for the main muscle groups of the extremities. In the plan, lumbopelvic, scapulothoracic and craniocervical neuromuscular efficiency exercises will also be included.
  Interventions: Other: Therapeutic exercise
- Control (Active Comparator): Get the training in with high-intensity interval exercise. Will be applied through 10 sets of 60 seconds. The first 30 seconds will consist of going up and down a step 15 cm high, immediately 30 seconds of squats as fast as possible with 90° knee flexion. The recovery period between each set will be 60 seconds, with a low-intensity activity (light walking). Based on high-intensity exercise, we must achieve an effort greater than 85% of the maximum frequency, using the heart rate meter and its equivalences with the Perceived Effort Scale (RPE).
  Interventions: Other: Therapeutic exercise

INTERVENTIONS:
Other: Therapeutic exercise — The control group and the experimental group will receive the training with high-intensity interval exercise. For a period of 12 weeks both groups will participate in their exercise program, which will be supervised by the physiotherapist in charge of the study; different from the one who will carry out the randomization and the one who will perform the evaluations. Women will attend 3 times a week for an hour to the "Hospital de especialidades" to receive their exercise program in which they participated. Both groups will receive therapeutic education to encourage adherence and self-management, which include aspects such as flexibility, musculoskeletal pain, physical performance, quality of life focused on physical and mental health, etc.
  Other Names: Physiotherapy

SUMMARY:
About 382 million of adults in the world have Diabetes type 2 (DT2), and it is foreseen that this number will increase to 592 million in 2035. International Diabetes Federation (IDF) (2017) established that 352 million adults around 20 and 79 years old (which is 7,3% of that population), could be classified as prediabetes. This last is characterized by the resistance to insulin of skeletal muscle, of the liver and/ or adipose tissue, provoking the excessive e insulin secretion of β cells and pancreatic exhaustion which produce severe hyperglycemia. The High-intensity interval training (HIIT) can increase the oxidation ability, relating directly to insulin sensibility.

DETAILED DESCRIPTION:
According to the latest research of the International Diabetes Federation (IDF) (2017), 352 million of adults around 20 and 79 years old (which is 7,3% of that population), could be classified as prediabetes. It is foreseen that this number will increase to 481 million in 2040. People with prediabetes have approximately 30% of the possibility to develop diabetes mellitus type 2 (DM2) during a term of 10 years. Prediabetes is characterized by levels of glucose in blood above the normal, but levels under the diagnostic standards of diabetes type 2. Prediabetes is an intermediate phase of hyperglycemia, even though there is no general agreement about the beginning of its determination. The American diabetes Association (ADA) said that it is characterized by glucose on disturbed fast (100-125 mg/dl), tolerance to disturbed glucose (140-199 mg/dl) and/or glycosylated hemoglobin, (HbA1c) which is around 5,7% and 6,4%. The World Health Organization (WHO) indicates that the beginning of prediabetes in glucose in fast is 110-125 mg/dl2. The etiology of prediabetes is mainly the resistance to insulin of skeletal muscle, the liver and / or adipose tissue which, and by the time, promotes excessive insulin secretion of B cells and produces a pancreatic exhaustion that produces severe hyperglycemia. The resistance to insulin of skeletal muscle is the essential responsible for the intolerance to glucose (IGT, postprandial glucose at 2 h> 140 mg/dl). On the other hand, the resistance to hepatic insulin is shown mainly as an alteration of glucose in fast (IFG; plasma glucose in fast >100 mg/dl), this last, because the production of glucose is excessive despite normal insulinemia. There are several research which prove that diabetes has a relation cause-effect with cardiovascular illness and mortality in all vascular causes. However, it is not an unavoidable process but reversible.

Even though it is probable that prediabetes will be the result of multiple factors, the deteriorated mitochondrial function is the main factor that contributes to the etiology of resistance to insulin, a crucial sign of this illness. The intervention designed to increase oxidative capacity in adults with diabetes, therefore, could relieve resistance to insulin and improve tolerance to glucose. Physical exercise is a vital known strategy to prevent, care and control diabetes type 2 and prediabetes.

Energy deficit after high intensity exercise contributes to increasing the sensibility of insulin. In fact, an Energy deficit of about 6,5 kcal/kg of corporal weight after a series of severe exercise resulted in an increase of the area under the curve (AUC) of postprandial insulin about 22% lower during an oral glucose tolerance test (OGTT). This last, in comparison with a reduction of 11% when there is a replacement of expended calories. This suggests that approximately 50% of the effect of the exercise to insulin sensibility is the result of energy deficit because of the exercise.

The high-intensity interval training (HIIT) can increase the oxidative capacity in comparison to continuous training in healthy individuals, which suggests the variation in fat oxidation depends on the intensity. This last observation is clinically relevant since fat oxidation during exercise is directly related to insulin sensitivity. The changes included for the HIIT in the mitochondrial function can explain its greater efficiency to provoke positive metabolic adaptations in comparison with traditional training treatment protocols of resistance, even when there is no diet intervention test to lose weight. Interval training (HIIT), training with corporal weight, and functional training has emerged as some attractive options to program therapeutic exercise in the ambit of physiotherapy. This is used as a systematic way and safe in different populations, including people at chronic illness risk.

Excess weight (body mass index (BMI) ≥ 25.0 kg/m2) and obesity (BMI ≥ 30.0 kg/m2) are common contributors to pain and disability in the musculoskeletal system, especially in the female population. Excessive weight increases mechanical stress on the joints and tissues of the body and cause physical limitations and body pain. It is evident an increase of pain severity in higher body mass index (BMI) ratings. With 40% of women worldwide classified as overweight and 15% as obese, the relation between pain and BMI may evolve as a growing challenge for the health system. The evidence suggests that obesity modulates pain through several mechanisms, such as mechanical load, inflammation, and psychological state. Obesity has been associated with markers of chronic inflammation, such as C-reactive protein levels, tumor necrosis factor α, amyloid A and interleukin 6 and white blood cell counts. Therefore, the impact of obesity on various musculoskeletal conditions may be due not only to the biomechanical stress of obesity, but also to the systemic effects. The latter suggests that increased inflammation caused by obesity may play a role in pain. The increased fat index and decreased muscle mass have been significantly associated with musculoskeletal pain among women, having higher rates of physical inactivity. Pain in obesity contributes to the deterioration of physical capacity, health-related quality of life and functional dependence.

The research has shown that pain limits participation in physical activity in general. Overweight and obese women have reported that fear of pain or injury during exercise is a major barrier to a more active lifestyle, as well as an important impediment to exercise adherence. However, physical activity, and especially resistance training, can prevent or reverse pain symptoms by increasing muscle mass, muscle strength, and physical function, helping stabilize joints, improve mobility, and improve proprioception. While acute exercise can transiently exacerbate pain symptoms, regular participation in exercise can reduce the severity or prevalence of pain. Also, while published attrition rates with regular exercise are high (around 50%), exercise adherence can be improved with exercise modifications, including accumulating several sets of exercise rather than one long session, which reduces the joint's range of motion and replaces impact with non-impact activity. Regular exercise has been identified as the primary prevention against more than 35 chronic conditions, including obesity, conditions related to joint pain, anxiety, and depression. Exercise stimulation can have a positive impact on chronic pain mediators by exerting anti-inflammatory effects, increasing muscle strength and coordination, and improving psychological outlook. A study conducted to evaluate the impact of a musculoskeletal pain intervention before participating in a weight management program; the Physiotherapy intervention aimed at decreasing musculoskeletal pain in obese individuals reported that musculoskeletal pain was reduced for those who completed the program. Given these findings, it is plausible that activity deterrence is a problem in this population. In contrast, specialized musculoskeletal interventions have been shown to reduce pain and improve exercise compliance even in chronic conditions.

The improvements in physical ability could take place if the exercise program includes resistance training, to avoid poor outcomes with women's health. strength is closely related to changes in the neuromusculoskeletal system, as well as reduction in muscle mass. The inclusion of resistance exercise training in such programs can further increase performance, skeletal muscle mass, resting metabolic rate, and energy expenditure and thus improve body composition and overall health. Resistance exercise protocols that incorporate whole-body movements, which aim to activate the entire neuromuscular system, can also improve the functional ability to perform activities of daily living in people who demonstrate neuromuscular limitations and reduced mobility.

Further to these conditions, emerging evidence indicates that movement patterns that increase the risk of musculoskeletal alterations occur due to neuromuscular control deficits, which lead to compensatory motor strategies. This lack of motor control or deficit in neuromuscular function has been operationally defined as the neurological mechanisms underlying the unconscious activation of dynamic constraints that occur in preparation for and in response to joint movement. Clinically, these deficits in neuromuscular control manifest as deficits in postural control and altered peripheral muscle activation, which arises from changes in the central nervous system that adversely affect the control of the skeletal muscular system. A core abdominal muscle training program improves the biomechanics of the lower extremities and trunk. biomechanical patterns may be favorable for preventing exercise-related injuries.

Improving self-regulation skills is a critical component to physical activity interventions that aim to reduce the risk of diabetes and promote independent long-term adherence. This last is a scientific position statement by the American Heart Association and the American Diabetes Association. Within this framework, the efficacy of self-regulation is a belief that refers to the confidence to promulgate and carry out self-managing behaviors. It is critical for successful long-term participation in behaviors such as physical activity. The self-efficacy has been identified as a significant predictor of the adoption and maintenance of physical activity behavior, as a mediator of the effects of the intervention on physical activity and it has been identified as the most influential factor of behavior change within the literature on physical activity. In this way, fostering strong beliefs about social, physical, and self-assessment outcomes, through therapeutic education, have the potential to influence people's motivation to adhere to an exercise program in Physiotherapy.

Advocating for a lower volume of physical activity is of potential importance for exercise adherence, as "lack of time" is the most common cited perceived barrier to regular participation in exercise. Lack of local facilities for physical exercise, as well as the economic resources that are invested in this aspect, especially in developing countries are important obstacles for people to continue in training programs. Therefore, the recent alternative of HIIT protocols performed with body weight is gaining more and more strength.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with glycosylated hemoglobin HbA1c 39-47 mmol/mol (5.7% - 6.4%), according to the primary care registry, in the last 6 months 20,21,22.
* Women older than or equal to ≥30 to ≤60 years of age.
* To have a body mass index (BMI) greater than or equal to 25 kg/m2.
* Women who do not have any cognitive limitations to understand the information sheet and instructions, and freely sign the informed consent.

Exclusion Criteria:

* Uncontrolled medical problems include, but are not limited to, cardiovascular, pulmonary, rheumatological, hematological, oncological, infectious, neuromuscular, or psychiatric diseases; diabetes or another endocrine disease; immunosuppression.
* Current treatment with hormone therapy that may affect glucose metabolism.
* Current treatment with loop diuretics or thiazide diuretics.
* Current treatment with beta-blockers or peroral steroids.
* Bariatric surgery in the last 2 years.
* Women who present neuromusculoskeletal alterations that hinder or prevent the performance of the physical exercise.
* Alcohol/drug abuse at the time of inclusion.
* Pregnant or lactating women.
* Concomitant participation in another intervention study.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
The glycosylated hemoglobin A1c | 24 weeks
  To determine whether the exercise training program with intervals of high intensity, endurance and neuromuscular efficiency of large muscle groups decreases the level of glycosylated hemoglobin A1c to a greater extent than the high-intensity training program in prediabetic women, considering effective a decrease 0,17%

SECONDARY OUTCOMES:
The serum glucose level | 24 weeks
  To examine whether the exercise training program with intervals of high intensity, endurance and neuromuscular efficiency of large muscle groups, further decreases the serum glucose level, by means of laboratory tests, in prediabetic women, considering effective a decrease <100 mg/dl
The level of maximum oxygen consumption | 24 weeks
  To examine whether the exercise training program with intervals of high intensity, endurance, and neuromuscular efficiency of large muscle groups, increases to a greater extent the level of maximum oxygen consumption, by means of the modified Bruce stress test, in prediabetic women, considering an increase of 10% effective
The Visual Analog Scale | 24 weeks
  To examine whether the exercise training program with intervals of high intensity, endurance, and neuromuscular efficiency of large muscle groups, decreases the intensity of perceived pain, by means of the Visual Analog Scale, in prediabetic women, considering effective a decrease of 3 units

CONTACTS AND LOCATIONS:
Overall Officials: CLARA LUZ PEREZ QUIROGA, MCs, Principal Investigator — Universidad UPAEP
Locations (1):
- UPAEP, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Enhancing Exercise Responsiveness across Prediabetes Phenotypes by Targeting Insulin Sensitivity with Nutrition — https://pubmed.ncbi.nlm.nih.gov/29387730/
- See also: Effects of lifestyle changes on adults with prediabetes: A systematic review and meta-analysis — http://pubmed.ncbi.nlm.nih.gov/30076075/
- See also: Two Weeks of Interval Training Enhances Fat Oxidation during Exercise in Obese Adults with Prediabetes — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC6873115/
- See also: Effect of 12-Month Resistance Training on Changes in Abdominal Adipose Tissue and Metabolic Variables in Patients with Prediabetes: A Randomized Controlled Trial — http://pubmed.ncbi.nlm.nih.gov/31737686/
- See also: Management of prediabetes — http://pubmed.ncbi.nlm.nih.gov/29808066/
- See also: Prediabetes: Why Should We Care? — http://pubmed.ncbi.nlm.nih.gov/30788015/
- See also: High intensity, circuit-type integrated neuromuscular training alters energy balance and reduces body mass and fat in obese women: A 10-month training-detraining randomized controlled trial — http://pubmed.ncbi.nlm.nih.gov/30138475/
- See also: High-intensity interval neuromuscular training promotes exercise behavioral regulation, adherence and weight loss in inactive obese women — http://pubmed.ncbi.nlm.nih.gov/31478436/
- See also: Does low and heavy load resistance training affect musculoskeletal pain in overweight and obese women? Secondary analysis of a randomized controlled trial — http://pubmed.ncbi.nlm.nih.gov/30692018/
- See also: Relationships between body mass index, fat mass, muscle mass, and musculoskeletal pain in community residents — http://pubmed.ncbi.nlm.nih.gov/25185757/
- See also: Randomized trial assessing the impact of a musculoskeletal intervention for pain before participating in a weight management program — http://pubmed.ncbi.nlm.nih.gov/20040884/
- See also: Chronic pain management in the obese patient: a focused review of key challenges and potential exercise solutions — http://pubmed.ncbi.nlm.nih.gov/25709495/
- See also: Periodized and non-periodized resistance training programs on body composition and physical function of older women — http://pubmed.ncbi.nlm.nih.gov/30862526/
- See also: Time course of low- and high-volume strength training on neuromuscular adaptations and muscle quality in older women — http://pubmed.ncbi.nlm.nih.gov/24414336/
- See also: Eccentric Exercise to Enhance Neuromuscular Control — http://pubmed.ncbi.nlm.nih.gov/28571492/
- See also: Core-Muscle Training and Neuromuscular Control of the Lower Limb and Trunk — http://pubmed.ncbi.nlm.nih.gov/31386583/
- See also: High-Intensity Interval or Continuous Moderate Exercise: A 24-Week Pilot Trial — http://pubmed.ncbi.nlm.nih.gov/29762252/